CLINICAL TRIAL: NCT03881423
Title: Deep vs Moderate Neuromuscular Blockade on Surgical Conditions and Quality of Recovery in Day Case Laparoscopic Cholecystectomy
Brief Title: Deep vs Moderate Neuromuscular Blockade in Day Case Laparoscopic Cholecystectomy.
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Wahba bakhet (Other)
Collaborators: Elite medical center (Unknown)
Responsible Party: Sponsor-Investigator, Wahba bakhet, Lecturer, Ain Shams University
Organization: Ain Shams University (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: wbakhet
Record Dates: First submitted 2019-03-16; First posted 2019-03-19 (Actual); Last update posted 2019-10-29 (Actual); Status verified 2019-10

CONDITIONS: Muscle Relaxation
MeSH Terms: interventions — Rocuronium; Neuromuscular Blocking Agents

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Deep block (Active Comparator): In the deep NMB-group, a PTC of 1 to 2 twitches was maintained, and NMB was reversed with sugammadex at the end of surgery.
  Interventions: Drug: Rocuronium Bromide
- Moderate block (Active Comparator): In the moderate NMB group, a TOF count of 1 to 2 was maintained and NMB was reversed with a combination of neostigmine and glycopyrolate at the end of surgery.
  Interventions: Drug: Rocuronium Bromide

INTERVENTIONS:
Drug: Rocuronium Bromide — DEEP block to PTC 1-3
  Other Names: Neuromuscular blocker

SUMMARY:
Laparoscopic cholecystectomy (LC) is commonly performed on ambulatory basis as a result of its ability to improve postoperative quality of recovery (QOR) and significantly reduce hospital stay .

DETAILED DESCRIPTION:
Laparoscopic cholecystectomy (LC) is commonly performed on ambulatory basis as a result of its ability to improve postoperative quality of recovery (QOR) and significantly reduce hospital stay.

The surgeon requires a good surgical conditions to perform the operation, whereas the anesthesiologist is concerned with postoperative QOR. Pneumoperitoneium -associated expansion of the abdominal cavity during LC is related to postoperative pain.

and other physiological changes, affecting the postoperative QOR negatively . Poor postoperative QOR leads to prolonged hospital stay .

ELIGIBILITY:
Inclusion Criteria:

* ASA I and II

Exclusion Criteria:

* Neuromuscular disorders

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Surgical conditions | Intraoperative
  The surgeon assessed surgical condition every 10 minutes
Quality of recovery | 24 hours postoperative
  Quality of recovery-40 (QoR-40) questionnaire, which includes five general quality of life dimensions: physical independence (5 items), pain (7 items), .emotional state (9 items), psychological support (7 items), and physical independence (5 items). Each item was graded with a 5-point score: none of the time, some of the time,usually, most of the time and all of the time. The total score on the QoR- 40 questionnaire ranges from 40 to 200 representing, respectively, extremely poor to excellent

SECONDARY OUTCOMES:
Postoperative pain | During the length of hospital stay post surgery (on average 24 hours)
  Visual analogue scale with its 0 to 10 score range: (0 (no pain) to 10 ( Severe pain)

CONTACTS AND LOCATIONS:
Locations (1):
- Ainshams University Hospitals, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Sharing
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year
Access Criteria: Web